CLINICAL TRIAL: NCT04689334
Title: Surgical Residency Training Program in Somalia: Outcomes of 7 Years
Brief Title: General Surgery Residency Training in Low Income Countries
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Nuray COLAPKULU, MD, Istanbul Medeniyet University
Other Study IDs: SomaliaResidency
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Global Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Outcome — The number of surgeries

SUMMARY:
The general surgery residency program was initiated in 2013 between Istanbul Medeniyet University and Benadir University. A formal training program was established that covered 3-year theoretical and practical training that would form the structure of academic, clinical and technical criteria by evaluating all the requirements of the surgical residency training. A resident logbook was prepared to track exam results, practices, knowledge and skill status that the residents achieved in the training process. Candidates who graduated from medical school and were successful in the multiple-choice exam consisting of basic and clinical sciences were accepted to the program each year in different numbers according to the capacity. From the initiation, 16 surgeons -9 in 2016, 3 in 2017 and 4 in 2018- graduated from the program. This study was designed after the last resident group graduated and worked as an attending surgeon at least for a year.

DETAILED DESCRIPTION:
The data were collected from graduates who were working as surgeons in Somalia to reveal the features and numbers of elective, emergency, trauma, and non-general surgical interventions performed in a month. A questionnaire consisting of pathology, type and numbers of interventions performed in one month by graduate surgeons (GS), including general surgery and other specialties, was prepared.

ELIGIBILITY:
Inclusion Criteria:

1. surgeons who completed program
2. surgerons who currently working as an attending physician in Somalia

Exclusion Criteria:

1. surgeons who has not completed program
2. surgeons who did not completed the questionare

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 14 general surgeon who completed the program
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
number of surgical interventions in one month | 1 month
  quantitative

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided